CLINICAL TRIAL: NCT05405244
Title: A Multimodel Examination of Bromocriptine on Homeostatic and Hedonic Mechanisms of Food Intake in Individuals at High Risk for Type 2 Diabetes
Brief Title: Examination of Bromocriptine on Homeostatic and Hedonic Mechanisms of Food Intake in Individuals at High Risk for T2DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 16-3177; 1-17-JDF-031 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Results first posted 2022-08-10 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-05

CONDITIONS: Overweight and Obesity; Eating Behavior
Keywords: bromocriptine; dopamine agonist; TaqIA polymorphism; eating behavior; food intake; overweight; obesity
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior | interventions — Bromocriptine

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two possible intervention arms (active drug vs. placebo) at baseline. Following a 2-week washout period, participants receive the other intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bromocriptine, then Placebo (Other): During the first intervention visit, participants receive a single dose of 1.6mg of bromocriptine (2 0.8mg capsules). Following a 2-week washout period, participants return for the second intervention visit, where they receive 2 capsules of placebo (sugar free calcium supplement) matched in shape (circle) and color (white) to bromocriptine. Both bromocriptine and placebo are administered orally.
  Interventions: Drug: Placebo; Drug: Bromocriptine-QR
- Placebo, then Bromocriptine (Other): During the first intervention visit, participants receive 2 capsules of placebo (sugar free calcium supplement). Following a 2-week washout period, participants return for the second intervention visit, where they receive a single dose of 1.6mg of bromocriptine (2 0.8mg capsules). Both bromocriptine and placebo are administered orally.
  Interventions: Drug: Placebo; Drug: Bromocriptine-QR

INTERVENTIONS:
Drug: Placebo — 2 capsules, orally administered once
  Other Names: placebo (calcium supplement)
Drug: Bromocriptine-QR — 1.6mg (2 0.8mg capsules), orally administered once
  Other Names: quick-release (QR) bromocriptine (cycloset)

SUMMARY:
The current project applies an integrative three-prong approach to investigate the potential of the dopamine D2 receptor (DRD2) agonist bromocriptine to: 1) increase homeostatic satiation signaling, 2) alter neural circuitry to reduce hedonically motivated food intake, and 3) examines a genetic predisposition that may markedly impact the effectiveness of this medication in those at high risk for T2DM.

DETAILED DESCRIPTION:
Twenty-nine million Americans have diagnosed type 2 diabetes (T2DM), with fewer than half able to meet treatment goals and considerably more are at risk for development of T2DM. Implementation of healthy eating behavior has been identified as a barrier to T2DM treatment and efficacy. The determinants of eating behavior and weight regulation involve a complex interaction among individual-level homeostatic, hedonic, and genetic systems, and the external food environment. The high prevalence of obesity and T2DM suggests hedonic motivation to consume food overrides homeostatic satiation signaling, resulting in excess food intake. Elevated intake increases body mass and promotes T2DM incidence via dysregulation of glucagon-like peptide 1 (GLP-1), amylin, and adiponectin, which in turn can negatively impact T2DM treatment options.

Use of a pharmaceutical, such as bromocriptine, to aid in behavioral change is a novel method for treating and ameliorating T2DM and warrants investigation given that previous work has shown reward response to food images mediates T2DM control. Use of functional magnetic resonance imaging (fMRI) techniques to predict and evaluate hedonically-motivated eating behavior can be used to measure sensitivity to reward, and the role it plays in developing obesity, and is therefore an excellent tool to examine the associations among bromocriptine, satiety hormones, reward sensitivity and eating behavior.

Moreover, since 20-35% of the population carries the DRD2 TaqIA A1 allele, and 65% of the population is overweight or obese and at high risk for T2DM development or currently diagnosed, as much as 23% of the population may greatly benefit from dopamine agonist treatment. Despite the possibility that bromocriptine may have robust impact on T2DM treatment or as prevention therapy in those that are genetically predisposed, few data are available that directly examine the three systems (homeostatic, hedonic, genetic) available to assess whether a genetically-informed, personalized T2DM treatment is viable.

ELIGIBILITY:
Inclusion Criteria:

* Baseline BMI between 25 and 35

Exclusion Criteria:

* Individuals with current fMRI contraindications (e.g., metal implants, braces)
* Probable current Axis I psychopathology (e.g., major depression disorder, panic disorder, generalized anxiety disorder, bipolar disorder)
* Habitual use of cigarettes or illicit drugs
* Pregnancy or breastfeeding
* Diagnosis of serious medical problems (e.g., diabetes, cardiovascular disease, stroke)
* Current weight loss dieting and/or weight fluctuations great than 10 lbs in the previous 6 weeks
* Do not consume dairy
* Allergy to bromocriptine, dairy, and nuts

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle S Burger, MPH, RD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (Single 1-Day Visit)
Arm/Group | Bromocriptine, Then Placebo | Placebo, Then Bromocriptine
Started | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Bromocriptine, Then Placebo | Placebo, Then Bromocriptine
Started | 28 | 27
Completed | 24 | 26
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Second Intervention (Single 1-Day Visit)
Arm/Group | Bromocriptine, Then Placebo | Placebo, Then Bromocriptine
Started | 24 | 26
Completed | 24 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Cross-over design where participants receive either a single dose of bromocriptine or placebo at the initial visit. After a 2-week washout period, they receive the opposite drug at the cross-over visit.
Arm/Group | All Participants
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 31
  More than one race | 2
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Ad Libitum Food and Beverage Intake (g)
Description: Ad libitum food intake of highly-palatable snacks is assessed during each intervention arm. Participants are left alone for 25 minutes to eat as much as they want from a selection of snacks (M&Ms, Skittles, Doritos, cheddar popcorn) and a chocolate milkshake. Both snacks and milkshake are pre- and post-weighed to determine ad libitum food intake.
Time Frame: Within 15 minutes of completion of the ad libitum period
Population: Data was collected via an iPad and sometimes recorded no value, as such the decrease in the sample was due to missing data.
Measure: Mean (Standard Deviation); unit: g
Groups:
- Bromocriptine: All participants; post-bromocriptine administration
- Placebo: All participants; post-placebo administration
Arm/Group | Bromocriptine | Placebo
Number analyzed (Participants) | 47 | 47
g
  Snacks intake | 71.5 (58.5) | 81.9 (55.9)
  Milkshake intake | 24.9 (61.2) | 33.6 (66.1)
Statistical Analysis 1: Comparison: Bromocriptine vs Placebo; Snack intake; Test type: Superiority; p = 0.45, t-test, 2 sided
Statistical Analysis 2: Comparison: Bromocriptine vs Placebo; Milkshake intake; Test type: Superiority; p = 0.28, t-test, 2 sided

2. Primary Outcome: Hedonic Ratings of Food as Measured by a Visual Analog Scale
Description: Testing the effects of the drug on hedonic ratings (pleasantness, desire to consume) of milkshake and snacks on a scale from -100 to 100.
  Pleasantness was assessed by asking 'How pleasant is this taste?', with responses ranging from -100 (most unpleasant imaginable) to 100 (most pleasant imaginable).
  Desire to consume was assessed by asking 'How much would you want to eat/drink this?', with responses ranging from -100 (least desirable imaginable) to 100 (most desirable imaginable).
Time Frame: Up to 5 minutes prior to ad libitum period start
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bromocriptine | Placebo
Number analyzed (Participants) | 47 | 47
score on a scale
  Snack Pleasantness | 32.6 (15.8) | 32.2 (15.9)
  Snack Desire | 11.2 (22.4) | 14.6 (22.7)
  Milkshake Pleasantness | 22.7 (34.3) | 32.4 (15.5)
  Milkshake Desire | -5.1 (40.2) | -5.6 (41.2)
Statistical Analysis 1: Comparison: Bromocriptine vs Placebo; Pleasantness; Test type: Superiority; p = 0.89, t-test, 2 sided
Statistical Analysis 2: Comparison: Bromocriptine vs Placebo; Desire to consume; Test type: Superiority; p < 0.001, t-test, 2 sided

3. Primary Outcome: Change in Voxel-wise Blood Oxygen Level-Dependent (BOLD) Brain Activation in Response to Milkshake Anticipation and Receipt vs. Water
Description: The fMRI paradigm assesses evoked BOLD response to cue-elicited anticipation and receipt of a milkshake and water. A region-of-interest (ROI) approach is used to assess changes in BOLD signal in the striatum. The striatal response is assessed for the two contrasts of interest: milkshake>h2o anticipation and milkshake>h2o receipt. Positive values reflect a higher striatal BOLD activation for the milkshake; negative reflects a higher striatal BOLD activation for the water. Parameter estimates of the relative BOLD response to each of these contrasts are extracted and compared between the two arms.
  The paradigm has 64 trials and each trial starts with the presentation of a cue for 1s signaling the impending delivery of either 3 mL of highly palatable milkshake or a control water solution over a period of 6s. Taste delivery is followed by a wait period and rinse (tasteless solution). The next trial begins after a 1-9s jitter. Order of milkshake and water trials is pseudo-randomized.
Time Frame: Baseline and 2 Weeks
Population: Participants who had issues with neuroimaging data (e.g., excessive motion, errors with image registration) were excluded from the analysis. As such the decrease in sample is due to suboptimal quality fMRI data.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Bromocriptine | Placebo
Number analyzed (Participants) | 33 | 33
arbitrary units
  Milkshake cue > Water cue | 50.24 (180.43) | 15.66 (208.4)
  Milkshake taste > Water taste | -14.32 (57.68) | 3.75 (66.03)

4. Secondary Outcome: Ad Libitum Food and Milkshake Intake (g) by TaqIA Allele Status (A1 vs. A2/A2)
Description: Testing the drug by gene (TaqIA) interaction on ad libitum food intake (g).The presence of the high-risk A1 allele of the TaqIA polymorphism (rs1800497) in the DRD2 gene was determined from saliva samples and is compared to the A2/A2 variant.
Time Frame: Within 15 minutes of completion of the ad libitum period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Groups:
- Bromocriptine - TaqIA A1: Participants with the high risk TaqIA A1 allele; post-bromocriptine administration
- Bromocriptine - TaqIA A2/A2: Participants without the high risk TaqIA A1 allele; post-bromocriptine administration
- Placebo - TaqIA A1: Participants with the high risk TaqIA A1 allele; post-placebo administration
- Placebo - TaqIA A2/A2: Participants without the high risk TaqIA A1 allele; post-placebo administration
Arm/Group | Bromocriptine - TaqIA A1 | Bromocriptine - TaqIA A2/A2 | Placebo - TaqIA A1 | Placebo - TaqIA A2/A2
Number analyzed (Participants) | 28 | 19 | 28 | 19
g
  Snacks intake | 72.1 (64.3) | 70.7 (50.2) | 75.2 (46.1) | 91.4 (67.7)
  Milkshake intake | 26.1 (57.9) | 23.3 (67.2) | 35.5 (66.7) | 30.9 (67.1)

5. Secondary Outcome: Hedonic Ratings of Milkshake Pleasantness and Desire as Measured by a Visual Analog Scale by TaqIA Allele Status (A1 vs. A2/A2)
Description: Testing the drug by gene (TaqIA) interaction on hedonic ratings (pleasantness, desire to consume) of milkshake on a scale from -100 to 100. Testing the drug by gene (TaqIA) interaction on ad libitum milkshake (g). The presence of the high-risk A1 allele of the TaqIA polymorphism (rs1800497) in the DRD2 gene was determined from saliva samples and is compared to the A2/A2 variant.
  Pleasantness was assessed by asking 'How pleasant is this taste?', with responses ranging from -100 (most unpleasant imaginable) to 100 (most pleasant imaginable).
  Desire to consume was assessed by asking 'How much would you want to eat/drink this?', with responses ranging from -100 (least desirable imaginable) to 100 (most desirable imaginable).
Time Frame: Up to 5 minutes prior to ad libitum period start
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bromocriptine - TaqIA A1 | Bromocriptine - TaqIA A2/A2 | Placebo - TaqIA A1 | Placebo - TaqIA A2/A2
Number analyzed (Participants) | 28 | 19 | 28 | 19
score on a scale
  Pleasantness | 27.7 (2.5) | 15.1 (38.8) | 29.9 (29.7) | 12.2 (27.8)
  Desire | 3.7 (38.8) | -18.1 (40.3) | 16.6 (20.9) | -21.5 (36.2)

6. Secondary Outcome: Change in Voxel-wise Blood Oxygen Level-Dependent (BOLD) Brain Activation in Response to Milkshake Anticipation and Receipt vs. Water by TaqIA Allele Status (A1 vs. A2/A2)
Description: The fMRI paradigm assesses evoked BOLD response to cue-elicited anticipation and receipt of a milkshake and water. A region-of-interest (ROI) approach is used to assess changes in BOLD signal in the striatum. The striatal response is assessed for the two contrasts of interest: milkshake>h2o anticipation and milkshake>h2o receipt. Positive values reflect a higher striatal BOLD activation for the milkshake; negative reflects a higher striatal BOLD activation for the water. Parameter estimates of the relative BOLD response to these contrasts are extracted and used to test the drug by gene (TaqIA) interaction.
  The paradigm has 64 trials and each trial starts with the presentation of a cue signaling the impending delivery of either 3 mL of highly palatable milkshake or a control water solution over a 6s period. Taste delivery is followed by a wait period and rinse (tasteless solution). The next trial begins after a 1-9s jitter. Order of milkshake and water trials is pseudo-randomized.
Time Frame: Baseline and 2 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Bromocriptine - TaqIA A1 | Bromocriptine - TaqIA A2/A2 | Placebo - TaqIA A1 | Placebo - TaqIA A2/A2
Number analyzed (Participants) | 18 | 15 | 18 | 15
arbitrary units
  Milkshake cue > Water cue | 99.14 (139.86) | -8.44 (209.51) | 71.54 (176.11) | -51.4 (229.74)
  Milkshake taste > Water taste | -27.21 (41.91) | 1.16 (70.73) | -14.64 (45.95) | 25.82 (80.29)

ADVERSE EVENTS:
Time Frame: Following administration of initial study intervention at Visit 1 through completion of visit day and again starting with second intervention administration and continuing through study completion, a total of approximately 10 hours for both visits.
Groups:
- Bromocriptine: Single dose of bromocriptine 1.6mg (2 0.8mg capsules)
- Placebo: 2 capsules of placebo (sugar free calcium supplement) matched in shape (circle) and color (white) to bromocriptine
Arm/Group | Bromocriptine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/51
Other Adverse Events (participants affected / at risk) | 2/54 | 0/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bromocriptine (N=54) | Placebo (N=51)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT05405244/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT05405244/SAP_001.pdf